CLINICAL TRIAL: NCT04027517
Title: A Multi-center, Randomized, Open-label, Active-controlled, Parallel-group, Phase III Study to Compare the Efficacy and Safety of JTZ-951 With Darbepoetin Alfa in Anemic Patients With Chronic Kidney Disease Receiving Maintenance Hemodialysis.
Brief Title: A Study to Evaluate Efficacy and Safety of JTZ-951 Compared to Darbepoetin Alfa in Korean Renal Anemia Patients Receiving Hemodialysis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JWP-JTZ-301
Record Dates: First submitted 2019-07-10; First posted 2019-07-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2020-08

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — enarodustat; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JTZ-951 (Experimental): Oral doses once daily
  Interventions: Drug: JTZ-951
- Darbepoetin Alfa (Active Comparator): Intravenous doses of Darbepoetin Alfa administered once weekly
  Interventions: Drug: Darbepoetin Alfa

INTERVENTIONS:
Drug: JTZ-951 — Oral tablet
  * Dose adjustments as maintenance dose is allowed according to the result of Hb level.
  Other Names: enarodustat
  Arms: JTZ-951
Drug: Darbepoetin Alfa — Intravenous administration
  * Dose adjustments as maintenance dose is allowed according to the result of Hb level.
  Other Names: Nesp pre-filled syringe
  Arms: Darbepoetin Alfa

SUMMARY:
JTZ-951 is a currently being developed as a treatment for renal anemia. This study aims to evaluate the efficacy and safety of JTZ-951 following a switch from erythropoiesis-stimulating agent (ESA) in Korean subjects receiving HemoDialysis with renal anemia.

This study is a Phase III, open, active-controlled, parallel-group, multi-center study.

The total duration of the study will be 30 weeks including screening, treatment and follow-up.

DETAILED DESCRIPTION:
The primary objective is to demonstrate non-inferiority of JTZ-951 to darbepoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

1. Korean patients aged ≥ 19 years at the time of consent
2. Patients receiving hemodialysis (including hemodiafiltration) consistently three times a week for at least 12 weeks before Scr Visit 1
3. Patients with TSAT (Transferrin saturation) *2 > 20% or ferritin > 75 ng/mL at Scr Visit 1*1
4. Patients being treated with ESAs for as least 4 weeks before Scr Visit 1.
5. Patients receiving ESAs at protocol specified dose regimen (i.e., frequency and dose)
6. Patients who have received the same ESA received in most recent week before Scr Visit 1 as during the period between Scr Visit 1 and the day before Week 0 at the same total dose and dosing frequency a week*4.
7. Patients with pre-dialysis Hb levels measured after the maximum interdialytic interval at Scr Visit 1 and Scr Visit 2 (2 weeks after Scr Visit 1) of ≥ 9.5 g/dL and < 12.0 g/dL and a difference (in absolute value) between Scr Visit 1 and Scr Visit 2 of ≤1.0 g/dL

Exclusion Criteria:

1. Patients with poorly controlled hypertension
2. Patients with severe hepatobiliary disease
3. Patients with congestive heart failure (NYHA Class III or more) or unstable angina
4. Patients who have developed myocardial infarction, cerebral infarction (excluding asymptomatic cerebral infarction), or venous thromboembolism (pulmonary embolism or deep vein thrombosis) during the period between 24 weeks before Scr Visit 1 and Week 0.
5. Patients who will undergo an ophthalmological procedure (photocoagulation therapy or vitreous surgery) for the treatment of diabetic retinopathy, diabetic macular edema, or age- related macular degeneration during the period between Scr Visit 1 and the end of the study
6. Patients who have undergone erythrocyte transfusion during the period between 12 weeks before Scr Visit 1 and Week 0.
7. Patients who have received protein anabolic hormones, testosterone enanthate, or mepitiostane during the period between 12 weeks before Scr Visit 1 and Week 0.
8. Patients with severe hyperparathyroidism
9. Patients with severe infection, systemic blood disorder (e.g., myelodysplastic syndrome, aplastic anemia, abnormal hemoglobin disease), or hemolytic anemia, or patients with anemia caused by obvious bleeding lesions (e.g., gastrointestinal hemorrhage)
10. Patients who are suspected to have anemia caused by noninfectious chronic inflammatory disease (e.g., connective tissue disease)
11. Patients with malignancy (including hematological malignancy) or previous history of malignancy during the period between 5 years before Scr Visit 1 and Week 0
12. Patients with previous history of a serious drug allergy such as anaphylactic shock or a hypersensitivity to DA
13. Patients with current or previous history of drug dependence or alcohol dependence
14. Patients who have received another investigational product or have received treatment with an investigational device, or have participated in clinical research involving intervention (medical action beyond the scope of ordinary medical practice intended for research purposes) and received treatment within 12 weeks before Scr Visit 1
15. Patients who have previously participated in a clinical study of JTZ-951 and received the investigational product
16. Patients who are pregnant, lactating, or may be pregnant (the possibility of pregnancy cannot be ruled out by the PI or the SI based on the results of pregnancy test at Scr Visit 1)
17. Female patients of childbearing potential who have not agreed to use appropriate contraception methods (medically accepted contraceptive methods: surgical sterilization, intrauterine device, condom, diaphragm, etc.) from the time of signing of informed consent to the end of the study, or male patients who have not agreed to use appropriate contraception methods from the start of study treatment to the end of the study.
18. Other patients who, in the judgment of the PI or the SI, are ineligible for the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Difference in mean Hb level change during the evaluation period from baseline (evaluation period - baseline) between study arm and control arm | baseline and Week 20 to 24
  Hb level during the evaluation period is the mean of the Hb levels at Week 20, Week 22 and End of Treatment (Week 24 or at discontinuation).
Difference in mean Hb level between study arm and control arm during the evaluation period | baseline and Week 20 to 24
  Hb level during the evaluation period is the mean of the Hb levels at Week 20, Week 22 and End of Treatment (Week 24 or at discontinuation).

SECONDARY OUTCOMES:
Proportion of subjects with Hb level within the range of baseline ± 1.0 g/dL at Week 4 | Week4
Proportion of subjects with mean Hb level of ≥10.0 g/dL and <12.0 g/dL during the evaluation period | Week 20, 22, 24
Hb level at each Visit | Week 2, 4, 8, 12, 16, 20, 22, 24
Change from baseline in Hb level at each Visit | Week 0, 2, 4, 8, 12, 16, 20, 22, 24

CONTACTS AND LOCATIONS:
Overall Officials: Lee, Study Chair — JW Pharmaceutical
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278